CLINICAL TRIAL: NCT02996188
Title: Acute Hemodynamic Changes During Paracentesis
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Joachim Saur, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: IGR-paracentesis
Record Dates: First submitted 2016-12-14; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Tense Ascites; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with refractory tense ascites
  Interventions: Procedure: routine therapeutic paracentesis

INTERVENTIONS:
Procedure: routine therapeutic paracentesis

SUMMARY:
The aim of our study was to evaluate hemodynamic changes during routine paracentesis in tense ascites using non-invasive inert gas rebreathing.

ELIGIBILITY:
Inclusion Criteria:

* refractory tense ascites with indication for therapeutic paracentesis

Exclusion Criteria:

* pregnancy
* inability to give inform consent
* inability to perform rebreathing maneuver

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine therapeutic paracentesis due to refractory tense ascites at a university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
change in cardiac output | 30 minutes
  prior to and after paracentesis
change in systemic vascular resistance | 30 minutes
  prior to and after paracentesis

IPD SHARING:
Plan to Share IPD: No